CLINICAL TRIAL: NCT06606860
Title: A Placebo Controlled, Double-Blind, 3-Arm Phase I Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Doses of 20 mg/kg Oxantel Pamoate in Healthy Adult Volunteers
Brief Title: Safety, Tolerability and PK of Single and Multiple Doses of Oxantel Pamoate Tablets
Acronym: HELP-OXA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Ifakara Health Institute (Other); Drugs for Neglected Diseases initiative (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P1773-22A
Record Dates: First submitted 2024-09-12; First posted 2024-09-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Soil transmitted helminths; Phase I; Safety; Tolerability; Pharmacokinetics; Trichuriasis; Whipworm; Parasitic Diseases; Neglected Diseases
MeSH Terms: conditions — Trichuriasis; Parasitic Diseases; Neglected Diseases | interventions — oxantel pamoate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): Treatment with a single dose of 20 mg/kg oxantel pamoate followed by administration of two daily doses placebo
  Interventions: Drug: Oxantel Pamoate
- Arm 2 (Experimental): Treatment with three daily dose of 20 mg/kg oxantel pamoate
  Interventions: Drug: Oxantel Pamoate
- Arm 3 (Placebo Comparator): Treatment with three daily doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxantel Pamoate — Oxantel Pamoate tablet, 250mg
  Arms: Arm 1; Arm 2
Drug: Placebo — Placebo tablet
  Arms: Arm 3

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and pharmacokinetics of oxantel pamoate tablet after administration of a single and multiple dose in healthy male and female adult volunteers.

The main questions aim to answer if oxantel pamoate is safe and well tolerated in healthy volunteers and if is it absorbed by the human body.

A single dose and a multiple dose of oxantel pamoate will be compared to placebo to see if there are any different effects.

DETAILED DESCRIPTION:
Objectives:

Primary objective:

To investigate the safety and tolerability of oxantel pamoate after single and multiple oral administration of a chewable tablet formulation.

Secondary objective:

To investigate the pharmacokinetics (PK) of oxantel pamoate after single and multiple oral administration of a chewable tablet formulation.

Study Design:

This is a randomized, placebo controlled, double blind, 3-arm Phase I single centre study in a total of 45 healthy adults. The participants will be randomized into one of the following three study arms:

* Study arm 1, 20 participants: Treatment with single dose of 20 mg/kg oxantel pamoate on day 1 followed by administration of two daily doses placebo
* Study arm 2, 20 participants: Treatment with three daily dose of 20 mg/kg oxantel pamoate
* Study arm 3, 5 participants: Treatment with three daily dose of placebo PK sampling will be performed at 13 defined time points (baseline included).

The participants will be admitted to the ward one day prior to commencement of the study treatment (day -1) and will stay until one day after the last dose has been administered. They will have a final follow-up visit on day 14. The safety and tolerability will be assessed as of the first dosage up to the last follow-up visit. Biochemistry, haematology, coagulation and urinalysis will be checked at baseline, day 3 and at the final follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or non-pregnant (confirmed by a negative serum pregnancy test) and non-breastfeeding female participants, aged between 18 to 45 years at the time of consent.
* Written informed consent (IC) obtained before any study procedure.
* Ability to read and write and to understand the participant information sheet and the nature of the trial and any hazards from participating in it (following a test with a maximum of two attempts). Ability to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire trial.
* Women of childbearing potential (WOCBP) must agree to use a highly effective form of contraception from at least 28 days prior to first dosage to 30 days after discharge from the ward.
* Normal body weight range (BMI between 18 and 29.9 kg/ m2).

Exclusion Criteria:

* Participation in another clinical trial within 3 months prior to the study, or within 5-times the half-life of the drug tested in the previous clinical trial, whichever is longer (time calculated relative to the last dose in the previous clinical trial).
* Regular daily consumption of more than one liter of xanthine-containing beverages (e.g. tea, coffee, cola or chocolate drinks).
* Regular daily consumption of more than 5 cigarettes daily.
* Use of a prescription medicine during the 28 days before the first dose of trial medication or use of an over-the-counter medicine, during the 7 days before the first dose of trial medication.
* Use of dietary supplements or herbal remedies (such as St John's Wort) known to interfere with the CYP3A4 and/or P-gp metabolic pathway during the 28 days before the first dose of trial medication.
* Therapies which may impact on the interpretation of study results in the opinion of the Investigator.
* Medical, social condition, psychiatric disorder or occupational reasons that, in the judgment of the Investigator, is a contraindication to the protocol, may impair the volunteer's ability to give informed consent or effectively participate in the study, may significantly increase the risk to the volunteer because of participation in the study or may impair interpretation of the study data.
* Blood pressure (BP) and heart rate (HR) in supine position at the screening examination outside the ranges (systolic BP range: 105-136 mm Hg systolic, diastolic BP range: 58-84 mm Hg diastolic; HR range: 56- 96 beats/min).
* Febrile illness within 1 week before the start of study treatment.
* History of relevant diseases of vital organs, of the central nervous system or other organs.
* Known renal or hepatic impairment
* Participants with a history of allergies, non-allergic drug reactions, adverse reaction to any drug, or multiple drug allergies.
* Presence or history of drug or alcohol abuse in the last 10 years.
* Surgery (e.g. stomach bypass) or medical condition that might affect absorption of study drug taken orally.
* Clinically relevant abnormal medical history, concurrent medical condition, acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
* Relevant pathological abnormalities in the electrocardiogram (ECG) such as a second or third-degree AV block, prolongation of the QRS complex over 120 msec or of the QTcF-interval over 450 msec (corrected interval according to Fridericia's formula).
* Positive test for human immunodeficiency virus (HIV), hepatitis B or C.
* Positive stool or urine test for helminth infestation by Kato-Katz, urine filtration or Baermann test.
* Positive for malaria by thick blood smear (TBS).
* Presence of abnormal physical findings, or laboratory values at the screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
General safety (number, frequency, severity, seriousness and duration of adverse events) | After first dosage on day 0 to day 14
  Summarized statistics on adverse events will be reported under categories such as total adverse events, serious adverse events, treatment emerging adverse events
Heart rate from baseline | After first dosage on day 0 to day 14
  Change of pulse rate from baseline
Blood pressure from baseline | After first dosage on day 0 to day 14
  Change of blood pressure from baseline. Systolic and diastolic blood pressure will be assessed
Temperature from baseline | After first dosage on day 0 to day 14
  Change of axillary temperature from baseline
Respiratory rate from baseline | After first dosage on day 0 to day 14
  Change of respiratory rate from baseline
Creatinine value from baseline | After first dosage on day 0 to day 14
  Change of creatinine value from baseline
Alanine aminotransferase value from baseline | After first dosage on day 0 to day 14
  Change of alanine aminotransferase value from baseline
Aspartate aminotransferase value from baseline | After first dosage on day 0 to day 14
  Change of aspartate aminotransferase value from baseline
Total bilirubin value from baseline | After first dosage on day 0 to day 14
  Change of total bilirubin value from baseline
Sodium value from baseline | After first dosage on day 0 to day 14
  Change of sodium value from baseline
Potassium value from baseline | After first dosage on day 0 to day 14
  Change of potassium value from baseline
Blood urea nitrogen value from baseline | After first dosage on day 0 to day 14
  Change of blood urea nitrogen value from baseline
Haemoglobin value from baseline | After first dosage on day 0 to day 14
  Change of haemoglobin value from baseline
Red blood cell count from baseline | After first dosage on day 0 to day 14
  Change of red blood cell count from baseline
Mean corpuscular volume from baseline | After first dosage on day 0 to day 14
  Change of mean corpuscular volume from baseline
Mean corpuscular haemoglobin value from baseline | After first dosage on day 0 to day 14
  Change of mean corpuscular haemoglobin value from baseline
Mean corpuscular haemoglobin concentration from baseline | After first dosage on day 0 to day 14
  Change of mean corpuscular haemoglobin concentration from baseline
Platelets value from baseline | After first dosage on day 0 to day 14
  Change of platelets value from baseline
White blood cell count from baseline | After first dosage on day 0 to day 14
  Change of white blood cell count from baseline
Neutrophils value from baseline | After first dosage on day 0 to day 14
  Change of neutrophils value from baseline
Lymphocytes value from baseline | After first dosage on day 0 to day 14
  Change of lymphocytes value from baseline
Monocytes value from baseline | After first dosage on day 0 to day 14
  Change of monocytes value from baseline
Eosinophils value from baseline | After first dosage on day 0 to day 14
  Change of eosinophils value from baseline
Basophils value from baseline | After first dosage on day 0 to day 14
  Change of basophils value from baseline
Prothrombin time from baseline | After first dosage on day 0 to day 14
  Change of prothrombin time value from baseline
Activated partial thromboplastin time from baseline | After first dosage on day 0 to day 14
  Change of activated partial thromboplastin time value from baseline
Protein in urine from baseline | After first dosage on day 0 to day 14
  Change of proteine in urine from baseline
Blood in urine from baseline | After first dosage on day 0 to day 14
  Change of blood in urine from baseline

SECONDARY OUTCOMES:
Cmax of oxantel pamoate | Plasma samples taken pre-dose -0.5 hours prior first dose, then 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after first dose and 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after third dose
  Peak Plasma Concentration (Cmax) of oxantel pamoate, if detectable
Tmax of oxantel pamoate | Plasma samples taken pre-dose -0.5 hours prior first dose, then 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after first dose and 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after third dose
  Time to reach Cmax (Tmax), in case of plasma concentration determined.
AUC of oxantel pamoate | Plasma samples taken pre-dose -0.5 hours, then 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after first dose and 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after third dose
  Area under the curve (AUC) of the plasma concentration determined.
AUC (0-t) of oxantel pamoate | Plasma samples taken pre-dose -0.5 hours prior first dose, then 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after first dose and 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after third dose
  Concentration from time zero to the last quantifiable concentration at time t, in case plasma concentration can be determined.
T1/2 of oxantel pamoate | Plasma samples taken pre-dose -0.5 hours prior first dose, then 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after first dose and 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after third dose
  The plasma elimination half-life, In case plasma concentration can be determined.
AUC (tau) of oxantel pamoate | Plasma samples taken pre-dose -0.5 hours prior first dose, then 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after first dose and 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after third dose
  The area under the plasma concentration curve over dosing interval, in case plasma concentration can be determined.
AUC (0-∞) of oxantel pamoate | Plasma samples taken pre-dose -0.5 hours prior first dose, then 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after first dose and 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours after third dose
  The AUC of the plasma concentration from time zero to infinity with extrapolation of the terminal phase, In case plasma concentration can be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Paris, MD, PhD, Study Director — Swiss Tropical & Public Health Institute; Jennifer Keiser, PhD, Study Chair — Swiss Tropical & Public Health Institute; Hussein Mbarak, MD, Principal Investigator — Ifakara Health Insitute, Tanzania
Locations (1):
- Ifakara Health Institute, Bagamoyo, Tanzania

IPD SHARING:
Plan to Share IPD: No